CLINICAL TRIAL: NCT01214837
Title: A Phase 3b, Randomized, Open-Label, Multi-Center Study to Evaluate the Safety and Immunogenicity of 2 or 3 Doses of MenACWY Conjugate Vaccine in Healthy Infants and the Effects of a Booster Dose of MenACWY Administered in the Second Year of Life.
Brief Title: Safety and Immunogenicity of 2 or 3 Doses of MenACWY Conjugate Vaccine in Healthy Infants and the Effects of a Booster Dose of MenACWY Administered in the Second Year of Life
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59_36
Record Dates: First submitted 2010-09-27; First posted 2010-10-05 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal; ACWY; Conjugate Vaccine; Meningitis; Infants; Persistence
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis | interventions — MenACWY-CRM vaccine

ARMS (3):
- MenACWY3 (Experimental): Subjects received a 2-dose primary series at 2 and 4 months of age and a toddler dose at 12 months of age.
  Interventions: Biological: MenACWY-CRM; Biological: Routine Vaccines
- MenACWY4 (Experimental): All the subjects received a 3-dose primary series at 2, 4 and 6 months of age and a toddler dose at 12 months of age. Approximately half of the subjects had serum collected at Month 3, and the remainder had serum collected at Month 4.
  Interventions: Biological: MenACWY-CRM; Biological: Routine Vaccines
- Routine Vaccines (Placebo Comparator): Subjects received routine vaccines only, including PCV-13, at 2, 4 and 6 months of age and a toddler dose at 12 months of age.
  Interventions: Biological: Routine Vaccines

INTERVENTIONS:
Biological: MenACWY-CRM — This group received a 3-dose primary series at 2, 4, and 6 months of age and a toddler dose at 12 months of age. Approximately half of the subjects had serum collected at Month 3, and the remainder had serum collected at Month 4.
  Arms: MenACWY4
Biological: MenACWY-CRM — This group received a 2-dose primary series at 2 and 4 months of age and a toddler dose at 12 months of age.
  Arms: MenACWY3
Biological: Routine Vaccines — Each 0.5 mL dose of the pneumococcal 13-valent conjugate vaccine (diphtheria CRM197 protein) is formulated to contain approximately 2.2 μg of each of Streptococcus pneumoniae serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F saccharides.

SUMMARY:
The purpose of this study was to assess immunogenicity of a 3-dose versus 4-dose infant vaccination schedule including kinetics of immune response in the early phases of the series.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both genders who are in generally good health will be eligible for this study. For infants to be enrolled, the parents/legal representatives need to provide written informed consent and to be available for all study visits.

Exclusion Criteria:

* Serious, acute, or chronic illnesses are reasons for exclusion.

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 751 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (35):
  - Birmingham, Alabama
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Huntington Beach, California
  - Madera, California
  - Nampa, Idaho
  - Cotton ONeil Clinical Research, Topeka, Kansas
  - Bardstown, Kentucky
  - Bluegrass Clinical Research (Bardstown Road), Louisville, Kentucky
  - Bluegrass Clinical Research (Brownsboro Park Blvd), Louisville, Kentucky
  - Springfield, Kentucky
  - Haughton, Louisiana
  - Shreveport, Louisiana
  - Niles, Michigan
  - Lincoln, Nebraska
  - Children's Physicians Dundee, Omaha, Nebraska
  - Creighton Univ, Omaha, Nebraska
  - Binghamton, New York
  - Johnson City, New York
  - Syracuse, New York
  - Dayton, Ohio
  - Huber Heights, Ohio
  - Kettering, Ohio
  - Tulsa, Oklahoma
  - Kingsport, Tennessee
  - Lebanon, Tennessee
  - San Antonio, Texas
  - Tomball, Texas
  - Layton, Utah
  - Salt Lake City, Utah
  - St. George, Utah
  - Richmond, Virginia
  - Rockwood Clinic P S, Spokane, Washington
- Canada (3):
  - Greater Sudbury, Ontario
  - Toronto, Ontario
  - Pierrefonds, Quebec

REFERENCES:
- [Derived] Block SL, Shepard J, Garfield H, Xie F, Han L, Dull PM, Smolenov I. Immunogenicity and Safety of a 3- and 4-dose Vaccination Series of a Meningococcal ACWY Conjugate Vaccine in Infants: Results of a Phase 3b, Randomized, Open-label Trial. Pediatr Infect Dis J. 2016 Feb;35(2):e48-59. doi: 10.1097/INF.0000000000000965. PMID 26479973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 3 sites in Canada and 37 sites in United States of America.
Pre-assignment Details: All the enrolled subjects were included in the trial.
Groups:
- MenACWY4: All subjects received a 3-dose primary series at 2, 4 and 6 months of age and a toddler dose at 12 months of age. Approximately half of the subjects had serum collected at Month 3, and the remainder had serum collected at Month 4.
- Routine Vaccines: Subjects received routine vaccines only, including pneumococcal 13-valent conjugate vaccine (PCV-13), at 2, 4, 6 and 12 months of age.
Period: Overall Study
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Started | 249 | 256 | 246
Completed | 195 | 192 | 184
Not Completed | 54 | 64 | 62
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Withdrawal by Subject | 27 | 36 | 28
Not completed — Lost to Follow-up | 20 | 15 | 21
Not completed — Inappropriate Enrolment | 0 | 1 | 2
Not completed — Administrative Reason | 2 | 6 | 4
Not completed — Protocol Violation | 3 | 1 | 5
Not completed — Unable to Classify | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled population- All subjects who had signed an informed consent, undergone screening procedure(s) and were randomized.
Groups:
- Routine Vaccines: Subjects received routine vaccines only, including PCV-13, at 2, 4, 6 and 12 months of age.
- Total: Total of all reporting groups
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines | Total
Number analyzed (Participants) | 249 | 256 | 246 | 751
Age, Continuous [Mean (Standard Deviation); unit: Days] | 66.4 (7.1) | 66.7 (7.4) | 66.7 (7.0) | 66.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 123 | 106 | 355
  Male | 123 | 133 | 140 | 396

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Serum Bactericidal Activity Using Human Complement (hSBA) ≥ 1:8 Against N. Meningitidis Serogroups A, C, W and Y Following a 4-dose Schedule of Men ACWY Vaccination.
Description: The immune response was assessed in terms of percentage of subjects with hSBA ≥ 1:8 against N. meningitidis serogroups A, C, W and Y following 4 doses of Men ACWY vaccine given to infants at 2, 4, 6 and 12 months of age.
Time Frame: 13 months of age
Population: Analysis was done on the Toddler Per Protocol Population (PPS) - all subjects who received all doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to unblinding through 13 month timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY4
Number analyzed (Participants) | 152
Percentage of subjects
  Serogroup A (N=141) | 96 [91 to 98]
  Serogroup C | 99 [95 to 100]
  Serogroup W (N=138) | 99 [96 to 100]
  Serogroup Y (N=146) | 99 [96 to 100]

2. Primary Outcome: Percentage of Subjects With hSBA ≥ 1:8 Against N. Meningitidis Serogroups A, C, W and Y Following 4-Dose and 3-Dose Schedule of Men ACWY Vaccination.
Description: The immune response was assessed in terms of percentage of subjects with hSBA ≥ 1:8 against N. meningitidis serogroups A, C, W and Y following 4 doses of Men ACWY vaccine given to infants at 2, 4,6 and 12 months of age and 3 doses of Men ACWY given to infants at 2, 4 and 12 months of age.
Time Frame: 13 months of age
Population: Analysis was done on Toddler PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- MenACWY4: Subjects received a 3-dose primary series at 2, 4 and 6 months of age and a toddler dose at 12 months of age. Approximately half of the subjects had serum collected at Month 3, and the remainder had serum collected at Month 4.
Arm/Group | MenACWY3 | MenACWY4
Number analyzed (Participants) | 160 | 152
Percentage of subjects
  Serogroup A (N=146,141) | 88 [82 to 93] | 96 [91 to 98]
  Serogroup C | 95 [90 to 98] | 99 [95 to 100]
  Serogroup W (N=153,138) | 99 [96 to 100] | 99 [96 to 100]
  Serogroup Y (N=154,146) | 100 [98 to 100] | 99 [96 to 100]
Statistical Analysis 1: Comparison: MenACWY3 vs MenACWY4; Non-inferiority of Men ACWY 3-dose series (doses at 2, 4 and 12 months) to 4-dose series (doses at 2, 4, 6 and 12 months of age) against serogroup A at 13 months of age; Test type: Non-Inferiority or Equivalence — Non-inferiority will be concluded if the lower limit of the two-sided 95% CI for the difference in percentage of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups C, W and Y between the 3-dose series and (minus) the 4-dose series, is greater than -10%; Miettinen and Nurminen method; Vaccine group difference = -7, 95% CI 2-sided [-14 to -1]
Statistical Analysis 2: Comparison: MenACWY3 vs MenACWY4; Non-inferiority of Men ACWY 3-dose series (doses at 2, 4 and 12 months) to 4-dose series (doses at 2, 4, 6 and 12 months of age) against serogroup C at 13 months of age; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -4, 95% CI 2-sided [-8 to 0]
Statistical Analysis 3: Comparison: MenACWY3 vs MenACWY4; Non-inferiority of Men ACWY 3-dose series (doses at 2, 4 and 12 months) to 4-dose series (doses at 2, 4, 6 and 12 months of age) against serogroup W at 13 months of age; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 4: Comparison: MenACWY3 vs MenACWY4; Non-inferiority of Men ACWY 3-dose series (doses at 2, 4 and 12 months) to 4-dose series (doses at 2, 4, 6 and 12 months of age) against serogroup Y at 13 months of age; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = 1, 95% CI 2-sided [-2 to 4]

3. Secondary Outcome: Percentage of Subjects With hSBA ≥1:8 Against N. Meningitidis Serogroups A, C, W and Y at Baseline (2 Months of Age) and at 3, 4, 5, and 7 Months of Age.
Description: Antibody levels were assessed in terms of percentage of subjects with hSBA ≥ 1:8 against N. meningitidis serogroups A, C, W and Y at baseline (2 months of age) and at 3, 4, 5 and 7 months of age.
Time Frame: Baseline (2 months of age), 3 months, 4 months , 5 months and 7 months of age
Population: Analysis was done on Infant PPS - all subjects who received all doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to unblinding, through the 7 month timepoint.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Number analyzed (Participants) | 185 | 176 | 187
Percentages of subjects
  Serogroup A (baseline; N=0,0,166) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 4 [1 to 8]
  Serogroup A (3 months; N=0,82,0) | NA [NA to NA] — Data was not collected at this timepoint | 9 [4 to 17] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup A (4 months; N=0,70,0) | NA [NA to NA] — Data was not collected at this timepoint | 4 [1 to 12] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup A (5 months; N=157,0,0) | 43 [35 to 51] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup A (7 months; N=169,157,171) | 23 [17 to 30] | 84 [77 to 89] | 1 [0.015 to 3]
  Serogroup C (baseline; N=0,0,167) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 9 [5 to 14]
  Serogroup C (3 months; N=0,85,0) | NA [NA to NA] — Data was not collected at this timepoint | 28 [19 to 39] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup C (4 months; N=0,70,0) | NA [NA to NA] — Data was not collected at this timepoint | 41 [30 to 54] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup C (5 months; N=170,0,0) | 86 [80 to 91] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup C (7 months) | 71 [64 to 78] | 95 [91 to 98] | 1 [0.014 to 3]
  Serogroup W (baseline; N=0,0,157) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 20 [14 to 28]
  Serogroup W (3 months; N=0,84,0) | NA [NA to NA] — Data was not collected at this timepoint | 15 [9 to 25] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup W (4 months; N=0,71,0) | NA [NA to NA] — Data was not collected at this timepoint | 35 [24 to 47] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup W (5 months; N=162,0,0) | 86 [80 to 91] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup W (7 months; N=179,162,181) | 74 [67 to 81] | 99 [96 to 100] | 1 [0.014 to 3]
  Serogroup Y (baseline; N=0,0,150) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 7 [4 to 13]
  Serogroup Y (3 months; N=0,80,0) | NA [NA to NA] — Data was not collected at this timepoint | 8 [3 to 16] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup Y (4 months; N=0,69,0) | NA [NA to NA] — Data was not collected at this timepoint | 7 [2 to 16] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup Y (5 months; N=152,0,0) | 67 [59 to 75] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup Y (7 months; N=170,163,173) | 48 [40 to 55] | 94 [90 to 97] | 0 [0 to 2]

4. Secondary Outcome: Geometric Mean hSBA Titers Against N Meningitis Serogroups A, C, W and Y at Baseline (2 Months of Age) and at 3, 4, 5, and 7 Months of Age.
Description: Antibody levels were assessed in terms of geometric mean titers (GMTs) against N. meningitidis serogroups A, C, W and Y at baseline (2 Months of Age) and at 3, 4, 5, and 7 Months of Age.
Time Frame: Baseline(2 months of age), 3 months, 4 months , 5 months and 7 months of age.
Population: Analysis was done on the Infant PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Number analyzed (Participants) | 185 | 176 | 187
Titers
  Serogroup A (baseline; N=0,0,166) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 2.18 [2.05 to 2.33]
  Serogroup A (3 months; N=0,82,0) | NA [NA to NA] — Data was not collected at this timepoint | 2.63 [2.2 to 3.15] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup A (4 months; N=0,70,0) | NA [NA to NA] — Data was not collected at this timepoint | 2.18 [2 to 2.37] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup A (5 months; N=157,0,0) | 7.09 [5.62 to 8.94] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup A (7 months; N=169,157,171) | 3.68 [3.17 to 4.29] | 28 [23 to 35] | 2.02 [1.98 to 2.06]
  Serogroup C (baseline; N=0,0,167) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 2.52 [2.28 to 2.78]
  Serogroup C (3 months; N=0,85,0) | NA [NA to NA] — Data was not collected at this timepoint | 4.79 [3.71 to 6.19] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup C (4 months; N=0,70,0) | NA [NA to NA] — Data was not collected at this timepoint | 6.44 [4.83 to 8.59] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup C (5 months; N=170,0,0) | 50 [39 to 64] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup C (7 months) | 17 [14 to 22] | 86 [70 to 104] | 2.03 [1.97 to 2.08]
  Serogroup W (baseline; N=0,0,157) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 3.32 [2.82 to 3.9]
  Serogroup W (3 months; N=0,84,0) | NA [NA to NA] — Data was not collected at this timepoint | 3 [2.48 to 3.61] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup W (4 months;N=0,71,0) | NA [NA to NA] — Data was not collected at this timepoint | 4.38 [3.42 to 5.61] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup W (5 months; N=162,0,0) | 55 [42 to 71] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup W (7 months; N=179,162,181) | 17 [14 to 21] | 90 [77 to 104] | 2.04 [1.96 to 2.11]
  Serogroup Y (baseline; N=0,0,150) | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint | 2.47 [2.25 to 2.7]
  Serogroup Y (3 months; N=0,80,0) | NA [NA to NA] — Data was not collected at this timepoint | 2.5 [2.14 to 2.93] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup Y (4 months; N=0,69,0) | NA [NA to NA] — Data was not collected at this timepoint | 2.46 [2.16 to 2.79] | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup Y (5 months; N=152,0,0) | 20 [15 to 26] | NA [NA to NA] — Data was not collected at this timepoint | NA [NA to NA] — Data was not collected at this timepoint
  Serogroup Y (7 months; N=170,163,173) | 7.56 [6.29 to 9.08] | 52 [43 to 64] | 2 [2 to 2]

5. Secondary Outcome: Percentage of Subjects With hSBA ≥1:8 Following 2 and 3 Infant Doses of MenACWY.
Description: Percentage of subjects with hSBA ≥1:8 against N meningitis serogroups A, C, W and Y was assessed following 2 and 3 infant doses of MenACWY as measured prior to the toddler dose at 12 months of age.
Time Frame: 12 months of age.
Population: Analysis was done on the Toddler PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY3 | MenACWY4
Number analyzed (Participants) | 149 | 147
Percentage of subjects
  Serogroup A (N=141,138) | 6 [2 to 11] | 22 [15 to 30]
  Serogroup C | 19 [13 to 27] | 48 [39 to 56]
  Serogroup W (N=149,142) | 33 [25 to 41] | 66 [58 to 74]
  Serogroup Y (N=145,139) | 25 [18 to 33] | 55 [47 to 64]

6. Secondary Outcome: Geometric Mean hSBA Titers Following 2 and 3 Infant Doses of MenACWY.
Description: The immune response was assessed in terms of GMTs against N. meningitidis serogroups A, C, W and Y following 2 and 3 infant doses of MenACWY as measured prior to the toddler dose at 12 months of age.
Time Frame: 12 months of age
Population: Analysis was done on the Toddler PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY3 | MenACWY4
Number analyzed (Participants) | 149 | 147
Titers
  Serogroup A (N=141,138) | 2.28 [2.09 to 2.49] | 3.65 [3.08 to 4.33]
  Serogroup C | 3.54 [2.99 to 4.17] | 8.55 [6.75 to 11]
  Serogroup W (N=149,142) | 5.41 [4.39 to 6.67] | 13 [11 to 16]
  Serogroup Y (N=145,139) | 3.82 [3.24 to 4.49] | 9.65 [7.79 to 12]

7. Secondary Outcome: GMTs at 13 Months of Age After Completion of 3- and 4-Dose Series of MenACWY.
Description: Immune response was assessed in terms of GMTs against N meningitis serogroups A, C, W and Y at 1 month after completion of a 3- and 4- dose series of MenACWY.
Time Frame: 13 months of age
Population: Analysis was done on the Toddler PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY3 | MenACWY4
Number analyzed (Participants) | 160 | 152
Titers
  Serogroup A (N=146,141) | 59 [45 to 77] | 94 [76 to 117]
  Serogroup C | 124 [99 to 156] | 160 [130 to 198]
  Serogroup W (N=153,138) | 248 [202 to 303] | 244 [195 to 305]
  Serogroup Y (N=154,146) | 212 [175 to 258] | 254 [203 to 318]

8. Secondary Outcome: Percentage of Subjects With 4-fold Increase in hSBA Titers Against N Meningitis Serogroups A, C, W and Y Between 12 and 13 Months of Age.
Description: The immune response was assessed in terms of percentage of subjects with 4-fold increase in hSBA titers between post and pre toddler dose against N meningitis serogroups A, C, W and Y, 1 month after completing a 3- or 4-dose series of MenACWY.
Time Frame: 13 months of age
Population: Analysis was done on the Toddler PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY3 | MenACWY4
Number analyzed (Participants) | 147 | 147
Percentage of subjects
  Serogroup A (N=127,129) | 88 [81 to 93] | 95 [90 to 98]
  Serogroup C | 93 [88 to 97] | 91 [85 to 95]
  Serogroup W (N=140,131) | 98 [94 to 100] | 90 [84 to 95]
  Serogroup Y (N=139,136) | 100 [97 to 100] | 96 [91 to 98]

9. Secondary Outcome: Effect of Concomitant Administration of 2 or 3 Doses of MenACWY on Immune Response to PCV-13 Antigens at 7 Months of Age.
Description: Percentage of subjects with IgG concentration ≥ 0.35 μg/mL against pneumococcal conjugate vaccine (PCV-13) antigens at 7 Months of age following concomitant administration of 2 or 3 doses of MenACWY with PCV-13.
Time Frame: 7 months of age.
Population: Analysis was done on the Infant PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Number analyzed (Participants) | 160 | 137 | 158
Percentage of subjects
  1 (N=159,136,156) | 93.7 [88.7 to 96.9] | 100 [97.3 to 100] | 94.2 [89.3 to 97.3]
  3 (N=150,129,147) | 79.3 [72 to 85.5] | 87.6 [80.6 to 92.7] | 82.3 [75.2 to 88.1]
  4 (N=160,137,157) | 94.4 [89.6 to 97.4] | 97.1 [92.7 to 99.2] | 96.8 [92.7 to 99]
  5 (N=156,133,154) | 84 [77.3 to 89.4] | 93.2 [87.5 to 96.9] | 88.3 [82.2 to 92.9]
  6A (N=159,136,156) | 98.1 [94.6 to 99.6] | 99.3 [96 to 100] | 98.1 [94.5 to 99.6]
  6B (N=160,137,157) | 84.4 [77.8 to 89.6] | 94.9 [89.8 to 97.9] | 84.7 [78.1 to 90]
  7F (N=158,136,156) | 100 [97.7 to 100] | 100 [97.3 to 100] | 99.4 [96.5 to 100]
  9V (N=159,136,157) | 89.3 [83.4 to 93.6] | 96.3 [91.6 to 98.8] | 92.4 [87 to 96]
  14 (N=158,136,158) | 99.4 [96.5 to 100] | 100 [97.3 to 100] | 97.5 [93.6 to 99.3]
  18C (N=158,136,157) | 97.5 [93.6 to 99.3] | 97.8 [93.7 to 99.5] | 100 [97.7 to 100]
  19A (N=158,135,156) | 95.6 [91.1 to 98.2] | 92.6 [86.8 to 96.4] | 98.1 [94.5 to 99.6]
  19F (N=159,136,158) | 100 [97.7 to 100] | 100 [97.3 to 100] | 99.4 [96.5 to 100]
  23F (N=158,136,158) | 93 [87.9 to 96.5] | 95.6 [90.6 to 98.4] | 91.1 [85.6 to 95.1]
Statistical Analysis 1: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 1; Test type: Non-Inferiority or Equivalence — Non-inferiority will be concluded if the lower limit of the two-sided 95% CI for the between group difference (MenACWY3 minus Routine) in percentage of subjects with IgG concentration ≥ 0.35 μg/mL against each pneumococcal anti-capsular polysaccharide is greater than -10%; Miettinen and Nurminen method; Vaccine group difference = -0.5, 95% CI 2-sided [-6.1 to 5]
Statistical Analysis 2: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 1; Test type: Non-Inferiority or Equivalence — Non-inferiority will be concluded if the lower limit of the two-sided 95% CI for the between group difference (MenACWY4 minus Routine) in percentage of subjects with IgG concentration ≥ 0.35 μg/mL against each pneumococcal anti-capsular polysaccharide is greater than -10%; Miettinen and Nurminen method; Vaccine group difference = 5.8, 95% CI 2-sided [3 to 10.5]
Statistical Analysis 3: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -3, 95% CI 2-sided [-11.9 to 6]
Statistical Analysis 4: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 5.3, 95% CI 2-sided [-3.3 to 13.7]
Statistical Analysis 5: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -2.4, 95% CI 2-sided [-7.5 to 2.3]
Statistical Analysis 6: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 0.3, 95% CI 2-sided [-4.4 to 4.7]
Statistical Analysis 7: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -4.3, 95% CI 2-sided [-12.1 to 3.4]
Statistical Analysis 8: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 4.9, 95% CI 2-sided [-1.9 to 11.8]
Statistical Analysis 9: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = 0.04, 95% CI 2-sided [-3.7 to 3.8]
Statistical Analysis 10: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 1.2, 95% CI 2-sided [-2.2 to 4.8]
Statistical Analysis 11: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -0.3, 95% CI 2-sided [-8.4 to 7.7]
Statistical Analysis 12: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 10.2, 95% CI 2-sided [3.4 to 17.2]
Statistical Analysis 13: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = 0.6, 95% CI 2-sided [-1.7 to 3.5]
Statistical Analysis 14: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 0.6, 95% CI 2-sided [-2.1 to 3.5]
Statistical Analysis 15: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -3.1, 95% CI 2-sided [-9.7 to 3.4]
Statistical Analysis 16: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 4, 95% CI 2-sided [-1.5 to 9.7]
Statistical Analysis 17: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; vaccine group difference = 1.9, 95% CI 2-sided [-1.2 to 5.7]
Statistical Analysis 18: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = 2.5, 95% CI 2-sided [-0.2 to 6.3]
Statistical Analysis 19: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -2.5, 95% CI 2-sided [-6.3 to -0.2]
Statistical Analysis 20: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = -2.2, 95% CI 2-sided [-6.2 to 0.2]
Statistical Analysis 21: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = -2.5, 95% CI 2-sided [-7.1 to 1.6]
Statistical Analysis 22: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = -5.5, 95% CI 2-sided [-11.3 to -0.9]
Statistical Analysis 23: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = 0.6, 95% CI 2-sided [-1.7 to 3.4]
Statistical Analysis 24: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 0.6, 95% CI 2-sided [-2.1 to 3.4]
Statistical Analysis 25: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 2 doses of MenACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Miettinen and Nurminen method; Vaccine group difference = 1.9, 95% CI 2-sided [-4.2 to 8.2]
Statistical Analysis 26: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 7 months of age for Serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 2]; Miettinen and Nurminen method; Vaccine group difference = 4.5, 95% CI 2-sided [-1.4 to 10.5]

10. Secondary Outcome: Effect of Concomitant Administration of 3 or 4 Doses of MenACWY on Immune Response to PCV-13 Antigens at 13 Months of Age.
Description: Geometric mean concentrations (GMCs) of antibodies against PCV-13 vaccine antigens at 13 months of age following concomitant administration of a 3- or 4-dose series of MenACWY with PCV-13.
Time Frame: 13 months of age.
Population: Analysis was done on the Toddler PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Number analyzed (Participants) | 147 | 117 | 124
µg/mL
  1 (N=145,116,123) | 2 [1.7 to 2.36] | 2.16 [1.83 to 2.56] | 2.14 [1.8 to 2.54]
  3 (N=139,113,118) | 0.88 [0.74 to 1.05] | 0.97 [0.81 to 1.15] | 0.77 [0.64 to 0.93]
  4 (N=146,117,123) | 1.19 [0.99 to 1.42] | 1.45 [1.21 to 1.75] | 1.53 [1.27 to 1.86]
  5 (N=140,114,117) | 1.29 [1.11 to 1.49] | 1.35 [1.16 to 1.57] | 1.26 [1.08 to 1.48]
  6A (N=146,117,124) | 6.89 [5.78 to 8.21] | 9.01 [7.52 to 11] | 8.16 [6.77 to 9.82]
  6B (N=147,117,124) | 4.29 [3.6 to 5.11] | 5.23 [4.36 to 6.27] | 5.04 [4.18 to 6.08]
  7F (N=147,116,123) | 3.96 [3.42 to 4.58] | 5.14 [4.41 to 5.98] | 4.95 [4.23 to 5.78]
  9V (N=146,117,123) | 1.37 [1.17 to 1.61] | 1.85 [1.56 to 2.18] | 1.73 [1.46 to 2.05]
  14 (N=147,117,124) | 7.76 [6.51 to 9.26] | 7.86 [6.55 to 9.43] | 7.54 [6.25 to 9.09]
  18C (N=146,116,123) | 1.52 [1.28 to 1.8] | 2.34 [1.96 to 2.79] | 2.13 [1.78 to 2.55]
  19A (N=144,114,124) | 5.51 [4.61 to 6.6] | 5.23 [4.34 to 6.3] | 5.39 [4.45 to 6.51]
  19F (N=147,117,124) | 5.79 [4.9 to 6.85] | 6.19 [5.21 to 7.35] | 5.8 [4.86 to 6.92]
  23F (N=147,117,124) | 4.21 [3.49 to 5.09] | 4.84 [3.98 to 5.89] | 5.44 [4.45 to 6.65]
Statistical Analysis 1: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 1; Test type: Non-Inferiority or Equivalence — Non-inferiority will be concluded if the lower limit of the two-sided 95% CI around the ratio of GMCs between groups (MenACWY3 to routine vaccines) is greater than 0.5; ANOVA; GMC ratio = 0.94, 95% CI 2-sided [0.77 to 1.13]
Statistical Analysis 2: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 1; Test type: Non-Inferiority or Equivalence — Non-inferiority will be concluded if the lower limit of the two-sided 95% CI around the ratio of GMCs between the groups (MenACWY4 to routine vaccines) is greater than 0.5; ANOVA; GMC ratio = 1.02, 95% CI 2-sided [0.83 to 1.25]
Statistical Analysis 3: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 1.14, 95% CI 2-sided [0.93 to 1.4]
Statistical Analysis 4: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.25, 95% CI 2-sided [1.01 to 1.55]
Statistical Analysis 5: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 0.77, 95% CI 2-sided [0.62 to 0.96]
Statistical Analysis 6: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 0.94, 95% CI 2-sided [0.75 to 1.18]
Statistical Analysis 7: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 1.02, 95% CI 2-sided [0.86 to 1.21]
Statistical Analysis 8: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.07, 95% CI 2-sided [0.89 to 1.29]
Statistical Analysis 9: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 0.85, 95% CI 2-sided [0.69 to 1.04]
Statistical Analysis 10: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.1, 95% CI 2-sided [0.88 to 1.37]
Statistical Analysis 11: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 0.85, 95% CI 2-sided [0.69 to 1.05]
Statistical Analysis 12: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.04, 95% CI 2-sided [0.83 to 1.3]
Statistical Analysis 13: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 0.8, 95% CI 2-sided [0.67 to 0.95]
Statistical Analysis 14: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.04, 95% CI 2-sided [0.87 to 1.25]
Statistical Analysis 15: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 0.79, 95% CI 2-sided [0.66 to 0.96]
Statistical Analysis 16: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.07, 95% CI 2-sided [0.87 to 1.31]
Statistical Analysis 17: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 1.03, 95% CI 2-sided [0.84 to 1.27]
Statistical Analysis 18: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.04, 95% CI 2-sided [0.83 to 1.3]
Statistical Analysis 19: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 0.72, 95% CI 2-sided [0.59 to 0.87]
Statistical Analysis 20: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.1, 95% CI 2-sided [0.89 to 1.36]
Statistical Analysis 21: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 1.02, 95% CI 2-sided [0.83 to 1.27]
Statistical Analysis 22: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 0.97, 95% CI 2-sided [0.77 to 1.21]
Statistical Analysis 23: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 1, 95% CI 2-sided [0.82 to 1.22]
Statistical Analysis 24: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 1.07, 95% CI 2-sided [0.86 to 1.32]
Statistical Analysis 25: Comparison: MenACWY3 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 3 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 1]; ANOVA; GMC ratio = 0.77, 95% CI 2-sided [0.62 to 0.97]
Statistical Analysis 26: Comparison: MenACWY4 vs Routine Vaccines; To demonstrate non-inferiority of immune response to PCV-13 antigens after concomitant administration of 4 doses of Men ACWY with routine vaccines including PCV-13, versus administration of routine vaccines only, at 13 months of age for Serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 10, analysis 2]; ANOVA; GMC ratio = 0.89, 95% CI 2-sided [0.7 to 1.13]

11. Secondary Outcome: Percentage Of Subjects Reporting at Least One Severe Systemic Solicited Adverse Event.
Description: Safety was assessed as the percentages of subjects who reported severe solicited systemic adverse events within 30 minutes through day 7 of MenACWY administration with concomitant vaccines vs. concomitant vaccines alone.
Time Frame: Within 7 days
Population: Analysis was done on the Solicited Safety Set - All subjects in the Exposed Set with solicited adverse event data
Measure: Number; unit: Percentage of subjects
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Number analyzed (Participants) | 238 | 240 | 230
Percentage of subjects | 18 | 21 | 18

12. Secondary Outcome: Number Of Subjects Reporting Solicited Local or Systemic Adverse Events.
Description: Safety was assessed as the number of subjects who reported solicited local or systemic adverse events between 6 hours and day 7 after administration of MenACWY with concomitant vaccines vs. concomitant vaccines alone.
Time Frame: Day 1 through Day 7
Population: Analysis was done on Solicited Safety Set - All subjects in the Exposed Set with solicited adverse event data
Measure: Number; unit: Subjects
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Number analyzed (Participants) | 238 | 239 | 229
Subjects
  Injection site erythema | 72 | 64 | 79
  Injection site induration | 60 | 40 | 74
  Tenderness | 117 | 127 | 126
  Change in eating habits (N=238,238,229) | 104 | 104 | 93
  Sleepiness | 153 | 147 | 149
  Persistent crying | 140 | 137 | 112
  Irritability | 173 | 171 | 152
  Vomiting | 68 | 52 | 54
  Diarrhea | 89 | 69 | 68
  Fever (≥38.0°C) | 55 | 52 | 41
  Rash | 23 | 19 | 18
  Use of analgesic/antipyretic | 162 | 173 | 153

13. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Any Vaccination.
Time Frame: 13 months of age
Population: Analysis was done on the Unsolicited Safety Set - All subjects in the Exposed Set with unsolicited adverse event data.
Measure: Number; unit: Subjects
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Number analyzed (Participants) | 242 | 252 | 239
Subjects
  Any AE | 219 | 220 | 209
  At least possibly related AEs | 24 | 32 | 10
  SAEs | 11 | 19 | 11
  Deaths | 0 | 0 | 1
  Medically attended AEs | 210 | 211 | 198
  AEs resulting in premature withdrawal | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: 13 months of age
Description: Solicited local and systemic and unsolicited AEs were assessed for 7 days postvaccination.
  AEs and SAEs were assessed throughout the study period.
  Out of a total of 751 subjects enrolled in the study, 733 (98%) subjects were exposed to at least 1 study vaccination and provided safety information.
Arm/Group | MenACWY3 | MenACWY4 | Routine Vaccines
Serious Adverse Events (participants affected / at risk) | 11/242 | 19/252 | 11/239
Other Adverse Events (participants affected / at risk) | 238/242 | 233/252 | 228/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY3 (N=242) | MenACWY4 (N=252) | Routine Vaccines (N=239)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Congenital megacolon (Congenital, familial and genetic disorders) | 0 | 0 | 1
Krabbe's disease (Congenital, familial and genetic disorders) | 1 | 0 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 2 | 2 | 4
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory synctial virus bronchiolitis (Infections and infestations) | 2 | 5 | 2
Staphylococcal abscess (Infections and infestations) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1 | 0
Breath holding (Psychiatric disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY3 (N=242) | MenACWY4 (N=252) | Routine Vaccines (N=239)
Ear pain (Ear and labyrinth disorders) | 13 | 10 | 9
Conjunctivitis (Eye disorders) | 42 | 25 | 40
Constipation (Gastrointestinal disorders) | 10 | 21 | 19
Diarrhea (Gastrointestinal disorders) | 103 | 78 | 80
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 14 | 27
Teething (Gastrointestinal disorders) | 15 | 13 | 19
Vomiting (Gastrointestinal disorders) | 76 | 68 | 67
Crying (General disorders) | 140 | 138 | 112
Injection site erythema (General disorders) | 87 | 80 | 89
Injection site induration (General disorders) | 65 | 45 | 79
Injection site pain (General disorders) | 137 | 140 | 138
Irritability (General disorders) | 181 | 179 | 157
Pyrexia (General disorders) | 88 | 87 | 69
Bronchiolitis (Infections and infestations) | 34 | 36 | 30
Bronchitis (Infections and infestations) | 8 | 19 | 17
Candida nappy rash (Infections and infestations) | 13 | 6 | 7
Croup Infectious (Infections and infestations) | 13 | 16 | 16
Gastroenteritis (Infections and infestations) | 22 | 18 | 27
Otitis media (Infections and infestations) | 94 | 77 | 89
Otitis media acute (Infections and infestations) | 23 | 19 | 16
Rhinitis (Infections and infestations) | 20 | 17 | 15
Sinusitis (Infections and infestations) | 9 | 17 | 7
Upper respiratory tract infection (Infections and infestations) | 105 | 107 | 106
Viral infection (Infections and infestations) | 38 | 32 | 30
Viral rash (Infections and infestations) | 10 | 10 | 13
Somnolence (Nervous system disorders) | 162 | 154 | 158
Eating disorder (Psychiatric disorders) | 104 | 104 | 93
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 32 | 37
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 | 18 | 14
Wheezing (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 16
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 10 | 11 | 14
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 38 | 31 | 22
Eczema (Skin and subcutaneous tissue disorders) | 16 | 19 | 20
Rash (Skin and subcutaneous tissue disorders) | 29 | 31 | 35
Candidiasis (Infections and infestations) | 14 | 20 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No